CLINICAL TRIAL: NCT06459388
Title: Effects of Stabilizing Reversal and Rhythmic Stabilization Versus Pelvic Proprioceptive Neuromuscular Facilitation on Trunk Control, Postural Stability and Mobility in Stroke Patients
Brief Title: Stabilizing Reversal and Rhythmic Stabilization vs Pelvic Proprioceptive Neuromuscular Facilitation in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0276
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stabilizing Reversals and Rhythmic Stabilization (Experimental): This group will receive stabilizing reversals and rhythmic reversals technique. The patient will perform 3 sets with 15 repetitions in each session, 5 days per week for 8 weeks
  Interventions: Other: Stabilizing Reversals and Rhythmic Stabilization
- Pelvic Proprioceptive Neuromuscular Facilitation (Experimental): This group will receive Pelvic PNF protocol. The treatment protocol will be followed 5 days a week for 8 weeks (i.e. 20 sessions) and each session will last for 30 minutes.
  Interventions: Other: Pelvic Proprioceptive Neuromuscular Facilitation

INTERVENTIONS:
Other: Stabilizing Reversals and Rhythmic Stabilization — 3 sets with 15 repetitions in each session, 5 days per week for 8 weeks.
  Arms: Stabilizing Reversals and Rhythmic Stabilization
Other: Pelvic Proprioceptive Neuromuscular Facilitation — The treatment protocol will be followed 5 days a week for 8 weeks (i.e. 20 sessions) and each session will last for 30 minutes.
  Arms: Pelvic Proprioceptive Neuromuscular Facilitation

SUMMARY:
The goal of this clinical trial is to compare the effects of stabilizing reversal and rhythmic stabilization versus pelvic proprioceptive neuromuscular facilitation on trunk control, postural stability and mobility in stroke patients. The main question it aims to answer is:

Is there any difference in effects of stabilizing reversal and rhythmic stabilization versus pelvic proprioceptive neuromuscular facilitation on trunk control, postural stability and mobility in stroke patients?

Researchers will compare stabilizing reversal and rhythmic stabilization to pelvic proprioceptive neuromuscular facilitation to see if there any difference in effects of stabilizing reversal and rhythmic stabilization versus pelvic proprioceptive neuromuscular facilitation on trunk control, postural stability and mobility in stroke patient.

Participants will be divided into two groups:

Group A will receive stabilizing reversals and rhythmic reversals technique. The patient will perform 3 sets with 15 repetitions in each session, 5 days per week for 8 weeks.

Group B will receive Pelvic PNF protocol. The treatment protocol will be followed 5 days a week for 8 weeks (i.e. 20 sessions) and each session will last for 30 minutes.

DETAILED DESCRIPTION:
It will be a randomized clinical trial study in which non-probability convenience sampling will be used. The sample size will be 50. The participants fulfilling the inclusion criteria will be divided randomly into two groups through computerized table generator method of randomization. Baseline assessment of both groups will be done before the execution of interventions. Group A will receive stabilizing reversal and rhythmic stabilization protocols for 5 days per week for 8 weeks. Group B will receive pelvic PNF protocol 5 days per week for 8 weeks. Trunk Impairment scale will be used to assess trunk control, Postural assessment Scale and Functional Reach Test will be used to assess postural stability and Performance Oriented Mobility Assessment will measure the mobility at the baseline, at 4 weeks and after the completion of intervention at 8 weeks to find out the outcome measures of the participants. The data will be analyzed using SPSS version 24. Normality of data will be assessed through Kolmogorov-smirnov test. Difference between preintervention, mid-intervention and post-intervention readings will be calculated using repeated measure ANOVA for parametric data. For non-parametric data Kruskal Wallis test will be used. For between group analysis Independent sample t test will be used for parametric data and Mann Whitney test will be used for non-parametric data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of ischemic stroke.
* Both genders of stroke patients.
* Age of stroke patients between 40-65 years.
* Duration of stroke less than 6 months.
* Participants should be able to understand and follow simple verbal commands (MMSE

  * 24).

Exclusion Criteria:

* Recurrent history of stroke.
* Recent history of any trauma.
* Musculoskeletal disorders such as low back pain, arthritis, degenerative diseases of the lower limbs affecting motor performance, spinal deformity and contractures.
* Spasticity (modified Ashworth scale grade ≥3) or flaccidity in lower limbs and upper limbs.
* PNF treatment given to the pelvic region within 6 weeks.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Trunk Impairment Scale | 0 week, 4th week, 8th week
  TIS assesses static and dynamic sitting balance and trunk coordination in a sitting position. On the static and dynamic sitting balance and coordination subscales the maximal scores that can be attained are 7, 10 and 6 points. The total score for TIS ranges between 0 for a minimal performance to 23 for a perfect performance. Test/retest and inter observer reliability for the TIS total score (ICC) - 0.96 and 0.99, respectively.
Postural Assessment Scale | 0 week, 4th week, 8th week
  Postural assessment scale assess and monitor postural control after stroke. It contains 12 four-level items of varying difficulty for assessing ability to maintain or change a given lying, sitting or standing posture. The PASS consists of 2 sections (maintaining posture and changing a posture) with a 4-point scale (0 indicating no performance and 3 indicating maximum performance) to describe each task. The total score ranges from 0 - 36.
Functional Reach Test | 0 week, 4th week, 8th week
  Functional Reach Test (FRT) is a clinical outcome measure and assessment tool for ascertaining dynamic balance in one simple task. Measurements are interpreted as: 10"/25 cm or greater Low risk of falls, 6"/15cm to 10"/25cm Risk of falling is 2x greater than normal, 6"/15cm or less Risk of falling is 4x greater than normal unwilling to reach Risk of falling is 8x greater than normal.
Performance Oriented Mobility Assessment | 0 week, 4th week, 8th week
  Performance oriented mobility assessment assesses a person's perception of balance and stability during activities of daily living and their fear of falling. The POMA test has a gait score and a balance score. It uses a 3-point ordinal scale of 0, 1 and 2. Gait is scored over 12 and balance is scored over 16 totaling 28. The lower the score on the POMA test, the higher the risk of falling. 25-28 = low fall risk, 19-24 = medium fall risk, < 19 = high fall risk.

CONTACTS AND LOCATIONS:
Overall Officials: Wajiha Shahid, Phd*, Principal Investigator — Riphah International University
Locations (1):
- Lahore General Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No